CLINICAL TRIAL: NCT04308967
Title: Effects of Balance Exercises on Central Sensitization in Patients With Knee Osteoarthritis
Brief Title: Central Sensitization in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Emre Tirasci, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 96/17
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Osteo Arthritis Knee; Central Sensitisation
Keywords: central sensitisation; osteoarthritis; balance exercises
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance exercises and information (Experimental): Balance exercises six weeks and three days in a week and information about central sensitisation.
  Interventions: Other: balance exercises
- Information (No Intervention): Information about central sensitisation.

INTERVENTIONS:
Other: balance exercises — Three-stage progressive balance exercises will be applied.
  Arms: Balance exercises and information

SUMMARY:
The stimuli that activate nociceptors cause the dorsal horn of the spinal cord neurons to be sensitive to low-intensive afferent stimuli by decreasing the excitation threshold in patients with osteoarthritis. Although painful stimuli disappear, this situation causes pain to continue and a decrease in quality of life. Therefore, central sensitization should be considered and treated in patients with osteoarthritis. Although various pharmacological and electrophysiological agents are used in the treatment of central sensitization, adequate efficacy is not provided in patients with osteoarthritis. The aim of this study is to investigate the effects of balance exercises on central sensitization in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with primary knee osteoarthritis according to American College of Rheumatology criteria,
* To be stage 2-3-4 knee osteoarthritis according to Kellgren Lawrence radiological staging,
* To be with a central sensitization score of over 40 according to the CSI,
* To be able to fill the scales and accept to participate in the study.

Exclusion Criteria:

* Being diagnosed with secondary osteoarthritis or inflammatory rheumatic disease,
* Having cognitive impairment,
* To have been treated with physiotherapy, with an intra articular injection or with a surgery from the knee within a maximum of six months
* Having various diseases that may adversely affect performing balance exercises,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | Before intervention, change in CSI scores at sixth week, change in CSI scores at 3 months.
  CSI consists of 2 parts as A and B. Part A contains 25 items associated with central sensitization symptoms, and the person is asked to score each item between 0 (never) and 4 (always) and total score ranges from 0-100. It is accepted that there is central sensitization in individuals over 40 points. Part B consists of 10 diseases. In this section, it is questioned whether she was diagnosed one or more of these 10 diseases. If any of these diseases exist, the person is excluded from the study.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Before intervention, change in BBS scores at sixth week, change in BBS scores at 3 months.
  In this scale, the patient is asked to perform 14 different activities. Every activity is scored between 0 (the worst)- 4 (the best) and a maximum of 56 points can be obtained.There is a correct proportion between the height of the score obtained and the balance.
Western Ontario ve McMaster University Osteoarthritis Index (WOMAC) | Before intervention, change in WOMAC scores at sixth week, change in WOMAC scores at 3 months.
  It consists of three sections as pain, stiffness and physical function and a total of 24 questions and scoring for each question as 0 = none, 1 = mild, 2 = medium, 3 = severe, 4 = very severe. Total WOMAC rate increases as pain, stiffness and physical function deterioration increase
Y Balance Test | Before intervention, change in Y balance test scores at sixth week, change in Y balance test scores at 3 months.
  Y Balance Test was used to assess the dynamic balance. This test is inexpensive and easy to transport which can be administered by therapists with different expertise and has been shown to have high reliability. In this test, patient exerts an effort to reach maximum distance in three different directions with the one leg while standing on the other leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Faculty of Medicine, Physical Medicine and Rehabilitation Clinic, Adana, Turkey (Türkiye)